CLINICAL TRIAL: NCT06039098
Title: Investigating the Relationship Between Intracranial Pressure and Cerebral Blood Flow Using Near-infrared Diffuse Correlation Spectroscopy
Brief Title: Investigating CBF and ICP Using DCS
Acronym: ICP-CBF
Status: Completed | Type: Observational
Sponsor: Queen Mary University of London (Other)
Collaborators: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 317751
Record Dates: First submitted 2023-09-08; First posted 2023-09-15 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Traumatic Brain Injury; Intracranial Hypertension
MeSH Terms: conditions — Brain Injuries, Traumatic; Intracranial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: Participants are patients who are undergoing invasive ICP and ABP measurement as part of their normal medical treatment.
  Interventions: Device: DCS

INTERVENTIONS:
Device: DCS — DCS monitoring of brain

SUMMARY:
We aim to acquire data using DCS on patients who are undergoing invasive ICP and ABP monitoring on ITU as part of their normal treatment.

Data will then be correlated to derive various parameters including CBF and BFI.

All interventions are entirely non-invasive.

DETAILED DESCRIPTION:
Cerebral Autoregulation (CA) is the complex process whereby the body maintains constant blood flow to the brain (cerebral blood flow, CBF) over a wide range of mean arterial pressures (MAP) in order to provide constant oxygenation and nutrition supply to cerebral tissue. By balancing blood and cerebrospinal fluid (CSF) pressures, CA dynamically stabilises cerebral perfusion pressure (CPP) and hence blood flow. Disordered CA may result in reduced oxygen and nutrient delivery to the brain tissue leading to hypoxic and ischaemic damage resulting in significant morbidity and mortality.

High intracranial pressure (ICP) is frequently associated with failing CA. Hence ICP is routinely monitored in patients suffering from traumatic brain injury (TBI) and other conditions which may result in CA failure. Raised ICP contributes to the majority of mortalities following severe TBI. All currently available ICP monitoring systems require insertion of an electrical or pneumatic transducer into the cranial cavity, usually sited within the brain parenchyma but occasionally into the subdural space (between the brain and the skull) or into the ventricles. This is currently only performed by neurosurgeons and carries a small but significant risk of haemorrhage or infection.

Non-invasive ICP and hence CA monitoring would eliminate the risk of complications, could be used by all healthcare professionals, would extend the use to outside a hospital settings and may extend the range of conditions to benefit from ICP monitoring.

This project pilots an approach to expand our understanding of the basic physiological interplay between intracranial pressure, arterial blood pressure, and cerebral blood flow in adult in-patients.

A recently-developed form of near-infrared (NIR) optical sensing known as Diffuse Correlation Spectroscopy (DCS) offers an opportunity to investigate cerebral blood flow at the bed-side continuously. DCS measures blood flow in the microvasculature of the brain by determining a blood flow index (BFi).

A similar technology based on near-infrared spectroscopy (NIRS), was recently successfully applied by the Chief Investigator in the same population in the same manner as in the current proposal (IRAS ID: 219476, approved by the East of England - Cambridge Central Research Ethics Committee (18/EE/0276) on 14/02/19). We therefore have extensive experience working with optical instruments in these patient groups.

In this proposal we will use a custom DCS research instrument. This research instrument is designed to measure microvascular cerebral blood flow for neuroscience and neurological research applications. While this device is a bespoke instrument, built with this study in mind, it is based on established research technologies and has been tested successfully in more than 20 healthy volunteers and in a range of quality-control experiments to date. It uses a forehead-mounted optical probe that contains near-infrared light sources that can illuminate the brain tissue non-invasively and continuously. The light's path within brain tissue is modulated by the flow of blood in the cerebral microvasculature and it is ultimately absorbed or backscattered. The backscattered light is collected at a different point within the probe.

The interplay between mean arterial blood (MAP) (measured by means of an intra-arterial catheter (part of normal medical care for patients on ITU) or a non-invasive finger-cuff) and ICP affects the morphology of the pulsatile flow in the cerebral microvascular, so the analysis of these signals in unison will help us better understand the relationship between ICP (which is measured clinically), MAP (which is measured clinically) and cerebral blood flow (which is not). This in turn could help support new research into head injury management, notably ICP-targeted treatment regimes. Ultimately this could lead to significant improvements in secondary injury-related mortality, length of hospital stay and reduced post-trauma disability. In addition the non-invasive nature of the monitor could extend the range of medical conditions that may benefit from ICP and CA monitoring including stroke, brain tumour surveillance, hydrocephalus, pre-hospital care of trauma patients, routine anaesthetic and ICU monitoring systems and screening of patients with headache in primary care.

In addition, if successfully developed, this technology is likely to be extremely relevant to low and middle income countries where access to neurosurgeons (and hence ICP monitoring) is extremely limited.

ELIGIBILITY:
Inclusion Criteria:

* Invasive monitoring of ICP and ABP as part of normal treatment

Exclusion Criteria:

* Not meeting inclusion criteria.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The largest demographic of patients undergoing ICP monitoring is trauma, therefore the study population is patients who have suffered TBI and are undergoing ICP monitoring on ITU.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2023-01-05 (Actual); Primary Completion 2023-08-20 (Actual); Study Completion 2023-08-20 (Actual)

PRIMARY OUTCOMES:
DCS signal acquisition | 12 months
  Successful acquisition of DCS signals from brain tissue

SECONDARY OUTCOMES:
Correlation of DCS signals with routine physiological data measurements | 10 months
  Correlation of DCS signals with routine physiological data measurements
ML approach to derive secondary parameters | 10 months
  Machine learning approach to derive additional parameters non-invasively

CONTACTS AND LOCATIONS:
Locations (1):
- Royal London Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with organizations / individuals upon reasonable request.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Once data have been acquired
Access Criteria: Upon reasonable request to be determined by the CI.